CLINICAL TRIAL: NCT01544075
Title: Efficacy of Pain Neurophysiology Education in Combination With Psychologic Inoculation in Chronic Whiplash Associated Disorders : a Double-blind Randomised Controlled Trial
Brief Title: Efficacy of Pain Neurophysiology Education in Combination With Psychologic Inoculation in Chronic Whiplash
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Jessica Van Oosterwijck, Dr., Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 143201112788
Record Dates: First submitted 2012-02-21; First posted 2012-03-05 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Pain, Chronic; Whiplash Injury
MeSH Terms: conditions — Chronic Pain; Whiplash Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PNE+PI (Experimental): The interventional group who will receive the experimental PNE+PI treatment.
  Interventions: Behavioral: Pain neurophysiology education (PNE) and psychologic inoculation (PI)
- NS (Active Comparator): The control group who will receive the neck school treatment.
  Interventions: Behavioral: Neck school (NS)

INTERVENTIONS:
Behavioral: Pain neurophysiology education (PNE) and psychologic inoculation (PI) — 3 sessions of PNE+PI are given which include education on pain neurophysiology and applying the PI technique for which subjects are asked to refute sentences which are read by the therapist.
  Arms: PNE+PI
Behavioral: Neck school (NS) — 3 sessions of NS which includes advice on posture, ergonomics and on performing activities.
  Arms: NS

SUMMARY:
With the present study the investigators wish to examine if reconceptualisation of pain, by educating chronic whiplash-associated disorders (CWAD) patients on the neurophysiology of pain, in combination with psychologic innoculation is able to influence maladaptive (pain) cognitions, pain (inhibition) and movement performance, and reduce symptoms.

DETAILED DESCRIPTION:
Results from a previous pilot study conducted by the same investigators suggest that intensive pain neurophysiology education (PNE) is able to increase pain thresholds and improve pain behavior and pain-free movement performance in patients with CWAD. However these results have not been confirmed in a randomized controlled trial.

In addition, it has been emphasized that PNE is not a standalone treatment and that future research should examine PNE in combination with other treatment modalities. Another treatment modality that challenges people's beliefs and barriers is psychological inoculation (PI). However, it has not yet been examined if PI could be a useful component in the rehabilitation of chronic pain patients.

ELIGIBILITY:
Inclusion Criteria:

* WAD grades I to II according to the Quebec Task Force criteria
* with chronic pain as result of a whiplash injury
* 18-65 years of age and with Dutch as their native language will be able to participate

Exclusion Criteria:

* other comorbidities or health issues that could explain the pain complaints
* < 18years > 65 years
* pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Change in pain pressure thresholds (conditioned pain modulation) | Measured prior to (baseline=day 1) and immediate following (=day 13) the treatment. Long term changes examined at 3 months follow-up.
  Measures over different locations on the body. Used as test stimulus while a conditioning stimulus is applied (conditioned pain modulation).

SECONDARY OUTCOMES:
Change in scores on the Neck Disability Index questionnaire | Measured prior to (baseline=day 1) and immediate following (=day 13) the treatment. Long term changes examined at 3 months follow-up.
  The NDI was developed in 1991 as a modification of the Oswestry Back Pain Index and was the first instrument designed to assess self-rated disability in patients with neck pain. The NDI is scored from 0 (good function) to 50(poor function), and the percentage of disability can be obtained when the score is multiplied by two. The NDI is a valid and reliable instrument sensitive to measure changes within a population of patients with neck pain.
Changes in the scores on the Neurophysiology of Pain Test Questionnaire | Measured prior to (baseline=day 1) and immediate following (=day 13) the treatment. Long term changes examined at 3 months follow-up.
  This is a questionnaire developed by Moseley et al. which assess the knwoledge of pain physiology in patients. A total score of 19 can be obtained when adding up one point for each item anwsered correctly.
Changes in scores on the Tampa Scale Kinesiophobia Questionnaire | Measured prior to (baseline=day 1) and immediate following (=day 13) the treatment. Long term changes examined at 3 months follow-up
  The TSK is a 17-item questionnaire that measures the fear of (re)injury due to movement [48]. Items are scored on a 4-point Likert scale, and a total score is calculated(1-4 for each item) after inversion of the individual scores of items 4, 8, 12, and 16. The total scores for the TSK range from 17 to 68.
Changes in scores on the Pain Catastrophizing Scale Questionnaire | Measured prior to (baseline=day 1) and immediate following (=day 13) the treatment. Long term changes examined at 3 months follow-up.
  This selfreported questionnaire measures catastrophic thinking about pain and consists of 13 items describing different thoughts and feelings that individuals may experience when experiencing pain. Items are scored on a 5-point scale, and one general score can be obtained for the degree of catastrophic thoughts about pain by adding up all individual item scores. This general score can be subdivided into three subscales: Helplessness, Magnification, and Rumination. Higher scores correspond to more severe catastrophic thoughts about pain.
Changes in score on the Pain Coping Inventory Questionnaire | Measured prior to (baseline=day 1) and immediate following (=day 13) the treatment. Long term changes examined at 3 months follow-up.
  The PCI consists of six scales (33 items) measuring cognitive and behavioral pain-coping strategies that represent two higher order pain coping dimensions: active(distraction, transformation, and reducing demands) and passive (resting, retreating, and worrying).
Changes in the Chronic Pain Self Efficacy Questionnaire | Measured prior to (baseline=day 1) and immediate following (=day 13) the treatment. Long term changes examined at 3 months follow-up.
  This is a questionnaire which can be used to measure self efficacy in chronic pain patients.
Changes in the scores on the Whiplash Associated Disorders Symptom list | Measured prior to (baseline=day 1) and immediate following (=day 13) the treatment. Long term changes examined at 3 months follow-up.
  This is a self-reported measure for assessing symptom severity in patients with WAD. The questionnaire is composed of the most reported WAD symptoms in the literature and some autonomic symptoms. Every symptom is presented by a visual analog scale (VAS) (100 mm), a method that is known for its validity and reliability.
Changes in scores on the Short Form 36 questionnaire | Measured prior to (baseline=day 1) and immediate following (=day 13) the treatment. Long term changes examined at 3 months follow-up.
  The SF-36 is a questionnaire to measure general health. Score reach from 0 to 100, and higher scores are obtained when havind a better general health.
Changes in range of movement and pain during the Brachial Plexus Provocation Test | Measured prior to (baseline=day 1) and immediate following (=day 13) the treatment. Long term changes examined at 3 months follow-up.
  Brachial Plexus Provocation Test is a neurodynamic test during which the range of elbow extension corresponding with the moment of "pain onset" and "submaximal pain" can be measured reliably, both in laboratory and clinical conditions. At the completion of the test, the subjects are asked to rate pain on a Visual Analogue Scale.
Changes in pain during the Neck Extension Test | Measured prior to (baseline=day 1) and immediate following (=day 13) the treatment. Long term changes examined at 3 months follow-up.
  The Neck Extension Test is used to diagnose sensory disturbances in patients with whiplash and is able to discriminate between subjects with symptoms after a whiplash injury and subjects without head or neck complaints. During cervical extension the patient's willingness to perform the movement is registered and the degree of pain experienced during the test performance is measured using a VAS.
Changes is force during the Cranio Cervical Flexion Test | Measured prior to (baseline=day 1) and immediate following (=day 13) the treatment. Long term changes examined at 3 months follow-up.
  This is a clinical test of the anatomical action of the deep cervical flexor muscles and evaluates neuromotor control. The features assessed are the activation and isometric endurance of the deep cervical flexors as well as their interaction with the superficial cervical flexors during the performance of five progressive stages of increasing craniocervical flexion range of motion. It is a low-load test performed in the supine position with the patient guided to each stage by feedback from a pressure sensor placed behind the neck.
Hospital Anxiety and Depression Scale | Baseline=day1
  This questionnaire wil be used in order to examine whether patients are depressed.
Impact of Events Scale | Baseline=day 1
  This questionnaire will be used in order to examine whether post traumatic stress disorder in present in the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jo Nijs, Phd Msc, Study Director — Vrije Universiteit Brussel
Locations (1):
- Artesis College Antwerp, Antwerp, Belgium

REFERENCES:
- [Background] Van Oosterwijck J, Nijs J, Meeus M, Truijen S, Craps J, Van den Keybus N, Paul L. Pain neurophysiology education improves cognitions, pain thresholds, and movement performance in people with chronic whiplash: a pilot study. J Rehabil Res Dev. 2011;48(1):43-58. doi: 10.1682/jrrd.2009.12.0206. PMID 21328162